CLINICAL TRIAL: NCT04109222
Title: Collection of Serum Samples From Children 6 Months to < 9 Years of Age Who Received Fluzone® Quadrivalent and Adults ≥ 65 Years of Age Who Received Fluzone® High-Dose, Influenza Vaccines, 2019-2020 Formulations
Brief Title: Collection of Serum Samples From Children and Older Adults Receiving the 2019-2020 Formulations of Fluzone® Quadrivalent and Fluzone® High-Dose Influenza Vaccines, Respectively
Acronym: GRC00097
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GRC00097; U1111-1225-1118 (Other: UTN)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Fluzone Quadrivalent Influenza vaccine: 6 to < 36 Months (Experimental): Participants aged 6 to <36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, no preservative (0.5-mL), 2019-2020 formulation
- Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 years (Experimental): Participants aged 3 to 9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, no preservative (0.5-mL), 2019-2020 formulation
- Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 years (Experimental): Participants aged >=65 years received a of 0.5-mL dose of Fluzone high-dose vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone High-Dose vaccine, 2019-2020 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, no preservative (0.5-mL), 2019-2020 formulation — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: Fluzone® Quadrivalent, No Preservative
  Arms: Group 1: Fluzone Quadrivalent Influenza vaccine: 6 to < 36 Months; Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 years
Biological: Fluzone High-Dose vaccine, 2019-2020 formulation — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Arms: Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 years

SUMMARY:
The primary objective of the study was to provide sera (collected from participants before vaccination [Blood Sample 1] and after final vaccination [Blood Sample 2]) to the Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.

DETAILED DESCRIPTION:
All participants received 1 intramuscular injection of the study vaccine associated with their assigned group at Visit 1. For participants 6 months to < 9 years of age for whom 2 doses of influenza vaccine are recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second intramuscular injection of Fluzone Quadrivalent vaccine was administered at Visit 2 (28 days after Visit 1).

Blood specimens were obtained from all participants prior to the first vaccination:

* At Visit 1 (Day 0) and 28 days following the final vaccination (Visit 2, if no study vaccine was administered at Visit 2; or Visit 3, if a second dose of study vaccine was administered at Visit 2), for participants 6 months to < 9 years of age (Group 1 and Group 2)
* At Visit 1 and 21 (window, 21-28) days post-vaccination (Visit 2), for participants greater than or equal to (>=) 65 years of age (Group 3) Serious Adverse Events (SAEs), suspected unexpected serious adverse reactions (SUSARs), or Adverse Event of Special Interests (AESIs) were collected from Visit 1 through Visit 2 for participants receiving 1 dose of study vaccine, and from Visit 1 through Visit 3 for participants receiving 2 doses of study vaccine.

Study duration per participant was approximately 28 days for participants 6 months to less than (<) 9 years of age, and 21 days for participants >= 65 years of age.

ELIGIBILITY:
Inclusion criteria :

An individual who fulfilled all of the following criteria were eligible for study enrollment:

* Aged 6 months to < 9 years or >= 65 years of age on the day of first study vaccination (study product administration).
* For participants 6 to < 12 months of age, born at full term of pregnancy (>= 37 weeks) and with a birth weight >= 5.5 pounds (2.5 kilograms).
* Informed consent form (ICF) had been signed and dated by participants >= 65 years of age.
* Assent form had been signed and dated by participants 7 to < 9 years of age, and ICF had been signed and dated by parent(s) or guardian(s) for participants 6 months to < 9 years of age.
* Participant and parent/guardian (of participants 6 months to < 9 years of age) were able to attend all scheduled visits and complied with all study procedures.

Exclusion criteria:

An individual who fulfilled any of the following criteria were excluded from study enrollment:

* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2019-2020 influenza season) with either study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the 3 months preceding planned inclusion.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the 6 months preceding planned inclusion; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to study vaccine or to a vaccine containing any of the same substances.
* Thrombocytopenia, which might be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature >= 100.4 degree (°) Fahrenheit [38.0 °Celsius]). A prospective participant were not included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) or in-laws of the Investigator or employee with direct involvement in the proposed study.
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participants if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- United States (2):
  - Investigational Site Number 8400002, Bardstown, Kentucky
  - Investigational Site Number 8400001, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: GRC00097 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25269&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 30 September 2019 to 7 October 2019 at 2 active sites in the United States.
Pre-assignment Details: A total of 90 participants were enrolled and vaccinated in the study.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months: Participants aged 6 to <36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP), a second dose was administered at Day 28.
- Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years: Participants aged >=65 years received a 0.5-mL dose of Fluzone high-dose vaccine intramuscularly at Day 0.
Period: Overall Study
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 Years | Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years
Started (Vaccinated participants.) | 30 | 30 | 30
Completed | 29 | 30 | 30
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled and vaccinated participants.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months: Participants aged 6 to <36 months received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
- Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years: Participants aged >=65 years received 1 dose of 0.5-mL Fluzone high-dose vaccine intramuscular injection at Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 Years | Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 0 | 60
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 30 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.86 (0.29) | 5.43 (1.45) | 71.83 (5.16) | 26.38 (32.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 16 | 47
  Male | 12 | 17 | 14 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 29 | 25 | 30 | 84
  More than one race | 1 | 3 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Aged 6 Months to < 9 Years Who Provided Serum Samples for Analysis: Groups 1 and 2
Description: Blood samples were collected from participants before first vaccination at Visit 1 (Day 0; pre-vaccination) and at Day 28 after final vaccination either at Visit 2 (Visit 1 + 28 days) for participants who received 1 dose of influenza vaccine; or at Visit 3 (Visit 2 + 28 days) for participants who received 2 doses of influenza vaccine as recommended by ACIP. Collected blood samples were provided to Center for Biologics Evaluation and Research (CBER) for further analysis by World Health Organization (WHO), Centers for Disease Control and Prevention (CDC), and Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 0; pre-vaccination) and 28 days post-final vaccination at Visit 2/Visit 3
Population: Analysis was performed on all vaccinated participants i.e. the participants who have received at least 1 dose of the study vaccine. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 Years
Number analyzed (Participants) | 28 | 30
Participants
  Visit 1 | 28 | 30
  Visit 2 | 22 | 28
  Visit 3 | 3 | 2

2. Primary Outcome: Number of Participants Aged >= 65 Years Who Provided Serum Samples for Analysis: Group 3
Description: Blood samples were collected from participants before vaccination at Visit 1 (Day 0; pre-vaccination) and 21 days after vaccination (Visit 2). Collected blood samples were provided to CBER for further analysis by WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 0; pre-vaccination) and 21 days post-vaccination (Visit 2)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years
Number analyzed (Participants) | 30
Participants
  Visit 1 | 30
  Visit 2 | 30

ADVERSE EVENTS:
Time Frame: Serious adverse events data were collected from Day 0 (post-vaccination) up to end of the study (i.e., up to Day 21 for adult participants [>= 65 years], Day 28 for child participants [6 to < 9 years] who had received 1 dose and Day 56 for participants who had received 2 doses).
Description: Non-serious adverse event data were not planned to be collected in this study. Analysis was performed on all enrolled and vaccinated participants.
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 Years | Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to < 36 Months (N=30) | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to < 9 Years (N=30) | Group 3: Fluzone High-Dose Influenza Vaccine: >= 65 Years (N=30)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04109222/Prot_SAP_000.pdf